CLINICAL TRIAL: NCT05886426
Title: Diagnostic Performance of Dynamic Four-dimensional Computed Tomography (4DCT) Compared to Arthroscopy for Analysing Distal Radioulnar Joint Instability
Brief Title: 4DCT Wrist Reference and DRUJ
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 114440
Record Dates: First submitted 2023-05-12; First posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Distal Radioulnar Joint Sprain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Reference study: Healthy participants (bilateral scans so 60 wrists) will be needed for the volunteer study to determine the visibility of the wrist joints (DRUJ, CMC-1 and MCP-1); acquire normal values and investigate the left right differences between the wrists
  Interventions: Diagnostic Test: 4DCT wrist and standard CT wrist
- Reliability study: Healthy participants (20 wrists) that underwent a 4DCT scan for the volunteer study will be needed to undergo a second unilateral scan to investigate the intra-patient test-retest reliability of the protocol
  Interventions: Diagnostic Test: 4DCT wrist and standard CT wrist
- DRUJ instability group: Patients with chronic unilateral wrist pain, in this study suspect for DRUJ instability, will be studied to evaluate the effect of TFCC injury on the wrist kinematics and evaluate the use of 4DCT for the diagnosis of TFCC injury
  Interventions: Diagnostic Test: 4DCT wrist and standard CT wrist

INTERVENTIONS:
Diagnostic Test: 4DCT wrist and standard CT wrist — Dynamic CT aquistion of wrist during movement and standard static wrist CT

SUMMARY:
The study will consist of 3 parts. First a reference study is performed with healthy volunteers to investigate the viability of 4DCT scanning of the wrist for evaluating wrist bones configurations and movements (translations and rotations) during a new set of wrist motions that have not been evaluated in our previous study focused on the scapholunate ligament (NL72518.091.19). The following will be evaluated: the visibility of the DRUJ, the carpal metacarpal 1 (CMC-1) joint and the metacarpal phalangeal 1 (MCP-1) joint during clinically relevant wrist movements. Besides, in this study the difference is evaluated between between the left right wrist within participants during wrist motion. In future clinical practice the uninjured wrist may be used as a reference for the injured wrist, determining the left right difference in healthy volunteers will show the robustness of this technique. Subsequently a reliability study is performed to investigate the intra-patient test-retest reliability of our 4DCT scanning protocol. Lastly a diagnostic clinical study is performed on patients with chronic wrist pain, suspect for DRUJ instability. The objective of the clinical study is to determine the sensitivity and specificity of the 4DCT scan (during a series of movements in which DRUJ instability is predicted to be best visible) in the diagnosis of DRUJ instability in comparison with arthroscopic findings (gold standard). If the 4DCT shows to have a sensitivity and specificity comparable to that of wrist arthroscop

DETAILED DESCRIPTION:
Single institution, a explorative volunteer study with participants followed by a prospective clinical study in the Radboud University Medical Center.

30 healthy participants will be included who have no medical history of wrist trauma, surgery or wrist complaints and in age range of 20-50 and; and 30 patients with chronic unilateral wrist pain suspect for DRUJ instability.

For the volunteer study all 30 healthy participants first undergo a bilateral 3D CT scan in neutral wrist position for usage of reference. The field of view of this scan includes all carpal bones and the two forearm bones. The scan technique is a Toshiba delivered application and CE certified. Subsequently, the forearms are placed in a supporting frame which minimizes lower-arm motion during 4DCT image acquisition. Prior to image acquisition, participants will undergo a training session on how to move their wrist according to the imaging protocol. A bilateral dynamic 4DCT scan is made while actively moving the wrists according to a protocoled cycle of movements. To reduce radiation exposure, the z-axis coverage is reduced to 12 cm in the 4DCT scan. Videos of the wrist movements are shown to the participant during image acquisition, which will help the participants to perform the movements at a constant pace. This will provide images with highest quality and will provide the source data considering carpal bone movements and function of ligaments during active wrist motions.

For the reliability study 20 of the participants included in the volunteer study will additively undergo an extra unilateral 4DCT scan at least 15 minutes after the bilateral 4DCT scan. Which wrist is scanned is decided by random selection. Except for the scanning being performed unilateral instead of bilateral the protocol is exactly the same as the 4DCT protocol as described above.

For this DRUJ instability study, a static 3D CT scan and a dynamic 4DCT scan of the both wrists of the patient suspect for DRUJ instability will be done after the X ray which is performed during standard clinical practice. The protocol is the same as described above in the volunteer study but the patients follow the DRUJ movement protocol with movements that are clinically relevant for DRUJ instability diagnosis.

The following radiographic signs will be evaluated: radioulnar angle; sigmoid notch to ulnar head joint distance; radioulnar ratio; radioulnar line distance; subluxation ratio; epicentre distance; radioulnar joint volume; ulnar variance and ulnar head to carpal bones joint distance [25] [26] [27] [30] [31].

ELIGIBILITY:
Inclusion Criteria:

* Between 18-50 years (healthy volunteer only)
* A 3D CT scan is required.
* Informed consent from both the healthy volunteer and patient.

Exclusion Criteria:

A participant who meets any of the following criteria will be excluded from participation in the volunteer study:

* < 18 year and > 50 years
* medical history of wrist: trauma, pain and/or surgery
* persons with limited wrist movements
* wrists with arthritis on plain radiograph or 3D CT scan
* pregnancy

A patient with suspicion of DRUJ instability who meets any of the following criteria will be excluded from participation in the clinical study:

* medical history of wrist fracture, known ligament lesion other than the TFCC and/or wrist surgery
* inability to undergo diagnostic arthroscopy
* wrists with arthritis on plain radiograph or 3D CT scan
* pregnancy

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: For the volunteer study, healthy volunteers between 18-50 years of age are included. For the clinical study, patients with unilateral chronic wrist pain suspected for DRUJ instability are included. Clinically suspect of DRUJ instability is based on the presence of a combination of the following: pain at the ulnar side of the wrist, context of wrist trauma or chronic overload; a positive piano key test and/or a positive DRUJ stress test and/or positive ballottement test.
  Participants with major joint stiffness or medical history of wrist surgery or fracture (radius, ulna or one of carpal bones) will not be included.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Primary study parameter Volunteer study | 3 months
  60 wrists of 30 healthy participants will be scanned and quantitative (e.g. in millimetres or degrees) automatic measurements of the 4DCT parameters will be performed.
Primary study parameter Reliability study | 3 months
  40 wrists of 20 participants will be used (of which 20 wrists have been scanned during the Volunteer study and 20 are rescanned during the reliability study) and quantitative (e.g. in millimeters or degrees) measurements of the 4DCT parameters will be performed automatically.
Primary study parameter prospective Clinical study (DRUJ instability) | 1 year
  4DCT parameter measurements will be compared to arthroscopically proven TFCC injuries (based on Palmar classification using unpaired student T-tests or Wilcoxon's tests, depending on the distribution. We will construct an univariate logistical regression model with as outcome a TFCC injury at arthroscopy or not, and as independent variables each one of the continuous 4DCT parameters separately, corrected for the same 4DCT parameter values of the asymptomatic contralateral wrist (and demographic parameters if proven to have a significant effect). From this, we can abstract ROC curves for different 4DCT parameters to estimate the sensitivity and specificity of these parameters.

SECONDARY OUTCOMES:
Volunteer study secondary outcome | 3 months
  Intraclass correlation coefficient (ICC) of the quantitative measurements will be calculated to assess the intra- and interobserver variability and left right similarity.
Secondary outcome reliability study | 3 months
  Test-retest reliability will be calculated with the coefficient of multiple correlation evaluating the similarity between the two motion patterns. The total waveform reliability present between test and retest will be evaluated using the root mean square deviation.
Comparison with atroscopy (DRUJ instability) | 1 year
  To investigate different grades of TFCC-injury on 4DCT we plan to construct a multinomial logistic regression model with the outcome variables being the different Palmer grades of TFCC injury and the independent variables the 4DCT parameters
Demographic variables | 1 year
  A multivariate linear regression analysis will be performed to analyze the effect of demographic variables (age and sex) on the 4DCT parameters measured.

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte van der Heijden, Dr., Principal Investigator — Radboud University Medical Center